CLINICAL TRIAL: NCT02748954
Title: Mood Management Effects of Brief Unsupported Internet Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i4Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-009- H
Record Dates: First submitted 2016-04-12; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Mood
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Thoughts. (Experimental): Increasing helpful thoughts consisted of two psychoeducational segments (i.e., thoughts affect emotions, and how to manage harmful thoughts), and a list of "helpful thoughts" that participants could choose to use to increase their mood for the next week
  Interventions: Behavioral: Thoughts
- Activities. (Experimental): Increasing activity level included a brief description of how activities affect mood. Participants were then asked to choose the activities they could use to improve their mood from an available list of "helpful activities"; users were also able to generate their own helpful activities. Participants were also presented with examples of unhelpful activities such as staying in bed and being isolated.
  Interventions: Behavioral: Activities.
- Assertiveness (Experimental): Increasing assertiveness, consisting of tips for communicating assertively, and an example of an assertive statement. Participants were asked to describe a recent conflict and apply the intervention's assertiveness techniques to address the conflict
  Interventions: Behavioral: Assertiveness.
- Sleep hygiene (Experimental): Increasing sleep hygiene included a description on how sleep can affect mood. Participants were also asked to select from a list of helpful sleep hygiene suggestions to be practiced within the next week such as, "Don't take naps during the day" and "Use the bed/bedroom for sleep or sex only".
  Interventions: Behavioral: Sleep hygiene
- Own Methods (Active Comparator): wherein participants were asked to identify four of their own personal strategies that have helped them improve their mood in the past.
  Interventions: Behavioral: Own Methods

INTERVENTIONS:
Behavioral: Thoughts — Thoughts. Increasing helpful thoughts consisted of two psychoeducational segments (i.e., thoughts affect emotions, and how to manage harmful thoughts), and a list of "helpful thoughts" that participants could choose to use to increase their mood for the next week.
  Arms: Thoughts.
Behavioral: Activities. — Increasing activity level included a brief description of how activities affect mood. Participants were then asked to choose the activities they could use to improve their mood from an available list of "helpful activities"; users were also able to generate their own helpful activities. Participants were also presented with examples of unhelpful activities such as staying in bed and being isolated
  Arms: Activities.
Behavioral: Assertiveness. — Increasing assertiveness, consisting of tips for communicating assertively, and an example of an assertive statement. Participants were asked to describe a recent conflict and apply the intervention's assertiveness techniques to address the conflict.
  Arms: Assertiveness
Behavioral: Sleep hygiene — Increasing sleep hygiene included a description on how sleep can affect mood. Participants were also asked to select from a list of helpful sleep hygiene suggestions to be practiced within the next week such as, "Don't take naps during the day" and "Use the bed/bedroom for sleep or sex only".
  Arms: Sleep hygiene
Behavioral: Own Methods — wherein participants were asked to identify four of their own personal strategies that have helped them improve their mood in the past.
  Arms: Own Methods

SUMMARY:
The main goal of this study was to compare the effect of a one-session unsupported Internet intervention on participants' clinical symptoms (depressive and anxiety symptoms) and related variables (mood, confidence and motivation).

DETAILED DESCRIPTION:
The main goal of this study was to compare the effect of a one-session unsupported Internet intervention on participants' clinical symptoms (depressive and anxiety symptoms) and related variables (mood, confidence and motivation).

Method: A total of 765 adults residing in the United States took part in a randomized controlled trial. Participants were randomly assigned to one of five brief plain text interventions lasting five to ten minutes. The interventions designed to address depressive symptoms were: Thoughts (increasing helpful thoughts), Activities (increasing activity level), Sleep Hygiene, Assertiveness (increasing assertiveness awareness), Own Methods (utilizing methods that were previously successful). They were followed-up one week after consenting.

ELIGIBILITY:
Inclusion Criteria:

- most be U.S. citizens

Exclusion Criteria:

- non-U.S. residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9; Kroenke & Spitzer, 2002) scores | Baseline - 1 week follow-up
  Which is a widely used 10-item measure that screens for a presence of a major depressive episode as well as assesses the severity of depressive symptomatology over a 2-week period.

SECONDARY OUTCOMES:
mood- Likert-type question | Baseline - 10 minutes after the intervention - 1 week follow-up
  How would you describe your mood in the last 2 weeks? and had responses ranging from 0 = Extremely Negative to 9 = Extremely Positive
Motivation - Likert-type question | Baseline - 10 minutes after the intervention - 1 week follow-up
  How motivated are you to do something to improve your mood? and had responses ranging from 0 = Extremely Negative to 9 = Extremely Positive
Confidence - Likert-type question | Baseline - 10 minutes after the intervention - 1 week follow-up
  How confident are you that you are able to do something to improve your mood?and had responses ranging from 0 = Extremely Negative to 9 = Extremely Positive
usefulness - Likert-type question | Baseline - 10 minutes after the intervention
  Before you see the ideas we will be sharing with you, how likely do you think they will be useful?" and had responses ranging from 0 = Very Unlikely to 6 = Very Likely.
7-item Generalized Anxiety Disorder questionnaire | Baseline - 1 week follow-up
  self-report questionnaire for measuring the level of generalized anxiety symptoms over a two-week period

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Muñoz, Ph.D, Principal Investigator — Palo Alto University

IPD SHARING:
Plan to Share IPD: No